CLINICAL TRIAL: NCT01589341
Title: Prognostic Impact of Segmental Chromosome Aberrations in Non MYCN Amplified Neuroblastomas in Different Age Groups
Brief Title: Studying Chromosomes in Samples From Younger Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL12B7; NCI-2012-01961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000732465 (Other: Clinical Trials.gov); COG-ANBL12B7 (Other: Children's Oncology Group)
Record Dates: First submitted 2012-04-29; First posted 2012-05-01 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative studies: Archived DNA samples are analyzed (laboratory biomarker analysis) for segmental chromosome aberrations by MLPA, a PCR-based technique. The following genomic regions are being studied: 1p, 1q, 3p, 4p, 7q, 9p, 11q, and 17q, as are the copy numbers of MYCN, NAG, DDX1, and ALK genes.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research studies chromosomes in samples from younger patients with neuroblastoma. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the impact on overall survival of patients with non-MYCN neuroblastoma below 18 months of age as compared to neuroblastoma patients above 18 months of age.

OUTLINE:

Archived DNA samples are analyzed for segmental chromosome aberrations by multiplex ligation-dependent probe amplification (MLPA), a polymerase chain reaction (PCR)-based technique. The following genomic regions are being studied: 1p, 1q, 3p, 4p, 7q, 9p, 11q, and 17q, as are the copy numbers of MYCN, NAG, DDX1, and ALK genes.

ELIGIBILITY:
Inclusion Criteria:

* Samples from neuroblastoma patients who, according to risk stratification, did not receive cytotoxic treatment and did never receive chemotherapy and are in complete response (CR) OR patients who, according to risk stratification, did not receive cytotoxic treatment initially, but had a localized or a systemic (stage Ms or M) relapse with or without following chemotherapy

  * Low-risk Children Oncology Group (COG) designation: no initial cytotoxic treatment, any stage, any age, any outcome
* DNA from untreated neuroblastoma tumor samples (from patients in the age group below and from patients in the age group above 1.5 years of age) available from the COG, Europe, Israel, and Japan
* No MYCN amplification
* No Schwann cell stroma-rich tumors
* No tumor cell content below 60%
* No DOT
* No patients diagnosed before 1997 and after 2005
* No lack of follow-up data
* See Disease Characteristics
* No initial cytotoxic treatment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Neuroblastoma patient samples
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of diagnosis to the date of death from any cause, assessed up to 5 years
  Estimated by the Kaplan-Meier method.

SECONDARY OUTCOMES:
Event-free survival (EFS) | From the date of diagnosis to the date of disease progression, death from any cause, or secondary neoplasm, assessed up to 5 years
  Estimated by the Kaplan-Meier method.
Incidence of metastatic relapses using cumulative incidences | Up to 5 years
  Grey's test and the model of Fine and Grey will be used for the evaluation of statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ambros, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States